CLINICAL TRIAL: NCT02565797
Title: A Point-of-care, Pragmatic Comparative Prevention-effectiveness Trial of DabirAIR Alternating Pressure Overlay System to Reduce Hospital-acquired Pressure Ulcers in the Peri-operative Setting.
Brief Title: Comparative Prevention-effectiveness Trial of DabirAIR Overlay System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dabir Surfaces Inc (Industry)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DOS-2015-CT01-1
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Pressure Ulcer
Keywords: Decubitus Ulcer, Peri-operative, support surface, alternating pressure, neurosurgery
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DabirAIR overlay-ORICU (Experimental): Patients scheduled for neurosurgical procedures will be placed over DabirAIR alternating pressure overlay (placed on top of standard of care support surface) in the operating room and in the post-op ICU.
  Interventions: Device: DabirAIR alternating pressure overlay
- DabirAIR overlay-OR (Experimental): Patients scheduled for neurosurgical procedures will be placed over DabirAIR alternating pressure overlay (placed on top of standard of care support surface) in the operating room alone and on standard of care support surface in the post-op ICU.
  Interventions: Device: DabirAIR alternating pressure overlay
- Control-SOC (No Intervention): Patients scheduled for neurosurgical procedures will be placed on standard of care support surface in the operating room and post-op ICU. Data will be abstracted through retrospective chart review.

INTERVENTIONS:
Device: DabirAIR alternating pressure overlay — DabirAIR alternating pressure overlay is a dynamic support surface that is placed on top a mattress. The DabirAIR overlay provides periodic pressure relief through the alternate inflation and deflation of air cells.
  Arms: DabirAIR overlay-OR; DabirAIR overlay-ORICU

SUMMARY:
Henry Ford Health System will evaluate the DabirAIR overlay system (DOS) for its effectiveness in preventing hospital acquired pressure ulcer (HAPU) in the peri-operative setting. The primary objective of the study is to compare the prevention-effectiveness (incidence rate of HAPU) between DOS (treatment group) vs facility specific standard of care pressure-relieving device(s) (control group) peri-operatively to discharge.

DETAILED DESCRIPTION:
Pressure ulcers (PUs) are localized skin or underlying tissue injury resulting from pressure or from pressure combined with shear or friction. In the United States, the annual treatment cost of PUs has been estimated at $11 billion and the cost to manage a single-full thickness PU is almost $70,000. According to Beckrich and Aronovitch, in the U.S., almost 25% of the approximately 1.6 million PUs that develop in acute care settings are acquired intra-operatively during surgeries that last more than three hours. The average estimated cost of treatment for the PUs in surgical patients is $750 million - $1.5 billion per year.

Surgical patients are at high risk for developing pressure ulcers due to the presence of many risk factors that are specific to intra-operative environment. Intra-operative factors that contribute to the development of pressure ulcers include patient weight, age, type of surgery, time on operating table longer than 2.5 hrs, anesthetic agents, extra-corporeal circulation, use of heating blanket and presence of vascular diseases.

The DabirAIR overlay system (DOS) is a semi-disposable, multi-patient use, alternating pressure (AP) overlay for surgical and medsurg bed applications. The system was developed as a new and innovative tool for surgeons and perioperative professionals alike to help reduce the risks of deep tissue injury and hospital-acquired pressure ulcers resulting from long surgical procedures in the OR.

Henry Ford Health System will evaluate the DabirAIR overlay system (DOS) for its effectiveness in preventing hospital acquired pressure ulcer (HAPU) in the peri-operative setting. The evaluation will be done in patients scheduled for neurosurgical procedures (surgical procedures typically last longer than 3 hours). The primary objective of the study is to compare the prevention-effectiveness (incidence rate of HAPU) between DOS (treatment group) vs facility specific standard of care pressure-relieving device(s) (control group) peri-operatively to discharge. About 400 patients in the treatment group will have their neurosurgical procedures while lying on the DOS in the operating room. Half of the patients from the treatment group will also be placed on the DOS in the post-op ICUs and recovery units. Retrospective chart reviews will be performed for 400 patients who had neurosurgical procedures while lying on the facility specific standard of care support surfaces in the operating room and post-op ICUs.

It is hypothesized that the treatment group will have lower rate of HAPU compared to the control group due to the pressure relief benefits offered by DOS. Prevention of HAPU will result in improved quality of life and clinical outcomes and cost savings to the healthcare facility.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects
* 18 years of age and older
* Pre-planned neurosurgical procedure lasting more than 2.5 hours

Exclusion Criteria:

* Emergent cases without adequate documentation
* Patients with pre-existing pressure ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2015-11; Primary Completion 2018-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Incidence rate of peri-operative hospital-acquired pressure ulcers (HAPU) | Peri-operative (up to 5 days from date of surgery)
  Investigate the comparative prevention-effectiveness (incidence rate of hospital-acquired pressure ulcers (HAPU)) between DOS (treatment) vs facility specific pressure-relieving device(s) (control) peri-operatively to discharge. The primary outcome of interest in this study is development of a first acquired pressure ulcer in the hospital after surgery to discharge. Pressure ulcers identified within 5 days from date of surgery will be associated with the surgical procedure.

SECONDARY OUTCOMES:
Adverse events related to use of DabirAIR overlay | Peri-operative (up to 5 days from date of surgery)
  Lack of adverse events related to use of DabirAIR overlay (during active use of overlay in OR and ICU/CCU). If any adverse events are reported, the causative factors for the adverse events will be analyzed and the adverse event will be grouped as study-device related or unrelated.
Cost-benefit of using DabirAIR | Peri-operative (up to 5 days from date of surgery)
  Demonstrate the cost-benefit (return-on-investment) of DOS from the perspective of the hospital financial system. The main outcome measure is net financial costs or benefits per patient length of stay (LOS). Direct medical costs attributed to resource utilization, prevention devices and wound care will be estimated during the LOS in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Siddiqui, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data

REFERENCES:
- [Background] Reddy M, Gill SS, Rochon PA. Preventing pressure ulcers: a systematic review. JAMA. 2006 Aug 23;296(8):974-84. doi: 10.1001/jama.296.8.974. PMID 16926357
- [Background] Aronovitch SA. Intraoperatively acquired pressure ulcer prevalence: a national study. J Wound Ostomy Continence Nurs. 1999 May;26(3):130-6. doi: 10.1016/s1071-5754(99)90030-x. PMID 10711122
- [Background] Feuchtinger J, Halfens RJ, Dassen T. Pressure ulcer risk factors in cardiac surgery: a review of the research literature. Heart Lung. 2005 Nov-Dec;34(6):375-85. doi: 10.1016/j.hrtlng.2005.04.004. PMID 16324956
- [Background] Pope R. Pressure sore formation in the operating theatre: 1. Br J Nurs. 1999 Feb 25-Mar 10;8(4):211-4, 216-7. doi: 10.12968/bjon.1999.8.4.6686. PMID 10347405
- [Background] Beckrich K, Aronovitch SA. Hospital-acquired pressure ulcers: a comparison of costs in medical vs. surgical patients. Nurs Econ. 1999 Sep-Oct;17(5):263-71. No abstract available. PMID 10711175
- [Background] Kemp MG, Keithley JK, Smith DW, Morreale B. Factors that contribute to pressure sores in surgical patients. Res Nurs Health. 1990 Oct;13(5):293-301. doi: 10.1002/nur.4770130505. PMID 2236652
- [Background] Hoshowsky VM, Schramm CA. Intraoperative pressure sore prevention: an analysis of bedding materials. Res Nurs Health. 1994 Oct;17(5):333-9. doi: 10.1002/nur.4770170504. PMID 8090944
- [Background] Defloor T, De Schuijmer JD. Preventing pressure ulcers: an evaluation of four operating-table mattresses. Appl Nurs Res. 2000 Aug;13(3):134-41. doi: 10.1053/apnr.2000.7653. PMID 10960997
- [Background] Tschannen D, Bates O, Talsma A, Guo Y. Patient-specific and surgical characteristics in the development of pressure ulcers. Am J Crit Care. 2012 Mar;21(2):116-25. doi: 10.4037/ajcc2012716. PMID 22381988